CLINICAL TRIAL: NCT06623500
Title: Prospective Cohort Study on Clinical Characteristics of Thyroid Cancer in Different Iodine Status Areas
Brief Title: Iodine Nutrition Status and Clinical Characteristics of Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Hai-qing Zhang, Chief physician, Shandong Provincial Hospital
Other Study IDs: ShandongPH 20240902
Record Dates: First submitted 2024-09-25; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Excessive iodine group: Residents with thyroid cancer who have lived in high iodine areas for a long time (5 years or more). According to the report of Shandong Institute of Endemic Disease Prevention and Control, three sub centers were selected in Excessive iodine group (Jining/Liaocheng/Heze).
  Interventions: Dietary Supplement: Iodine excess
- Suitable iodine group: Residents with thyroid cancer who have lived in suitable iodine areas for a long time (5 years or more). According to the report of Shandong Institute of Endemic Disease Prevention and Control, three sub centers were selected in suitable iodine (Jinan/Shenyang/Haerbin) areas.
  Interventions: Dietary Supplement: Iodine suitable

INTERVENTIONS:
Dietary Supplement: Iodine excess — Iodine excess areas: water iodine ≥100μg/L; or urinary iodine concentration (median urinary iodine levels in children aged 8-10 years old)≥300μg/L
  Groups: Excessive iodine group
Dietary Supplement: Iodine suitable — Iodine suitable areas：water iodine ≥40μg/L and ≤100μg/L; or urinary iodine concentration(median urinary iodine levels in children aged 8-10 years old) 100-199μg/L.
  Groups: Suitable iodine group

SUMMARY:
The effect of iodine nutritional status on thyroid cancer has been controversial for many years. We designed a prospective cohort study that recruiting patients in different iodine areas who underwent thyroid cancer surgery in branch hospitals from 2012 to 2019，and follow up their clinical outcomes. We aimed to analyse the relationship between regional iodine nutrition level and pathological types, clinical features, and prognosis of thyroid cancer.

DETAILED DESCRIPTION:
Three sub centers were selected in high iodine (Jining/Liaocheng/Heze) and moderate iodine (Jinan/Shenyang/Haerbin) areas respectively. Patients lived in the above-mentioned regions for at least 5 years and diagnosed as thyroid cancer and underwent thyroid surgery in branch hospitals from 2012 to 2019 were recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18~65 years old, gender not limited;
2. Living in the selected region for at least 5 years;
3. Patients who underwent thyroid surgery at various research centers were pathologically diagnosed with thyroid cancer;
4. The clinical data （general information、surgical scope 、pathological report、utrasonic report, etc ）of the case is complete.

Exclusion Criteria:

1. Diagnosed as other types of cancer or thyroid metastatic cancer;
2. There are serious comorbidities such as heart, liver, and kidney diseases present;
3. Unable to follow up on prognostic information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three sub centers were selected in high iodine (Jining/Liaocheng/Heze) and moderate iodine (Jinan/Shenyang/Haerbin) areas respectively. Patients lived in the above-mentioned regions at least for 5 years who was diagnosed as thyroid cancer and underwent thyroid surgery in branch hospitals from 2012 to 2019 were recruited.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with recurrence | from enrollment to the final follow-up at 5 years
  Recurrence: diagnosed as the same type of thyroid cancer again by pathology
Number of participants with distant metastasis | from enrollment to the final follow-up at 5 years
  Distant metastasis: Pathological confirmed thyroid cancer occurring outside the thyroid gland
All-cause mortality | from enrollment to the final follow-up at 5 years
  The ratio of the total number of deaths caused by various reasons during the research period to the number of participants

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No